CLINICAL TRIAL: NCT00142298
Title: An Open Label Trial of Telbivudine (LdT) in Adults With Chronic Hepatitis B Previously Treated in Idenix-Sponsored Telbivudine Studies
Brief Title: Telbivudine in Adults Previously Treated in Idenix-Sponsored Telbivudine Studies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDT600A2303; NV-02B-022 (Other: Idenix)
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Results first posted 2011-07-25 (Estimated); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine

ARMS (1):
- telbivudine (Experimental): telbivudine 600 mg p.o. daily for 104 weeks.
  Interventions: Drug: Telbivudine (LdT)

INTERVENTIONS:
Drug: Telbivudine (LdT) — Telbivudine was to be supplied as white to off-white, oval, bi-convex tablets for the 200 mg tablets and white to off-white ovaloid, slightly curved, beveled edges, film coated tablets for the 600 mg tablets. Study drug (600 mg) was to be self-administered by patients orally (p.o.) in a once daily regimen for 104 weeks; for study consistency, the daily dose had to be taken at the same time each day, with or without food.
  Other Names: Sebivo®/Tyzeka®; LdT600

SUMMARY:
This trial is being conducted as an open-label, extended-term study for patients with chronic hepatitis B who have previously completed an Idenix-sponsored trial with telbivudine.

DETAILED DESCRIPTION:
Patients from 6 feeder trials could be eligible to enter current study CLDT600A2303 ( NCT00142298) if they met inclusion/exclusion criteria. The feeder studies were as follows:

* CLDT600A2302 (NV-02B-007)(NCT00057265), the GLOBE study, was a Phase III, randomized, doubleblind,multi-center, 104-week, pivotal study of telbivudine vs. lamivudine in treatment of naïve patients with compensated chronic hepatitis B. CLDT600A2302/NV-02B-007 (NCT00057265) is hereafter referred to as study 2302.
* NV-02B-015 (NCT00131742) was a Phase III, randomized, double-blind, 104-week study comparing the efficacy and safety of telbivudine (600 mg/day) to lamivudine (100 mg/day) in treatment of naïve Chinese patients with compensated chronic hepatitis B. NV-02B-015 (NCT00131742) is hereafter referred to as study 015.
* CLDT600A2301 (NV-02B-011)(NCT00076336) was a Phase III, randomized double-blind, multi-center, 104-week, pivotal study of telbivudine (600 mg/day) vs. lamivudine (100 mg/day) in treatment-naïve adults with decompensated chronic hepatitis B. CLDT600A2301/NV-02B-011 (NCT00076336) is hereafter referred to as study 2301.
* NV-02B-010 (NCT00124241) was a Phase IIb, 104-week extension study of telbivudine, lamivudine or the combination of both agents in patients with chronic hepatitis B who had completed the core study NV-02B-003 (NCT00124241). NV-02B-010 (NCT00124241) is hereafter referred to as study 010.

NV-02B-003 (NCT00124241) was a Phase IIa, 52-week study of telbivudine, lamivudine or the combination of both agents in patients with HBeAg-positive chronic hepatitis B.

* CLDT600A2401 (NV-02B-018) (NCT00115245) was a Phase IIIb, randomized, open-label, multi-center,52-week study of telbivudine vs. adefovir dipivoxil for 24 weeks then a switch to telbivudine for another 28 weeks in treatment-naïve patients with compensated chronic hepatitis B. CLDT600A2401/NV-02B-018 (NCT00115245) is hereafter referred to as study 2401.
* CLDT600A2402 (NV-02B-019) (NCT00132652) was a Phase IIIb, randomized, open-label, multi-center, 52-week study of switching lamivudine to telbivudine vs. continued on lamivudine treatment in adults with compensated chronic hepatitis B who were previously treated with lamivudine for 3-12 months. CLDT600A2402/NV-02-019 (NCT00132652) is hereafter referred to as study 2402.

PATIENT GROUPS:

GROUP A: Patients with HBeAg (+) or HBeAg (-) compensated chronic hepatitis B who did not discontinue treatment in their previous study due to an efficacy response and required further treatment or who had met the criteria for discontinuation of treatment in their previous study due to efficacy, but were being maintained on study drug by the principal investigator. For patients treated with telbivudine who enrolled into Group A from studies 2302 and 015, the total telbivudine treatment time (starting from feeder study baseline to the end of the on-treatment period in study 2303) was 208 weeks. For patients treated with lamivudine in studies 2302/015 and enrolled into group A and for all patients in group A from studies 2401/2402/010, the total telbivudine treatment time was 104 weeks.

GROUP B: Patients with HBeAg (+) or HBeAg (-) decompensated chronic hepatitis B who did not discontinue treatment in their previous study due to an efficacy response and required further treatment. Patients treated with telbivudine in study 2301 were enrolled to group B and the total telbivudine treatment time (starting from feeder study baseline to the end of the on-treatment period in study 2303) was 208 weeks. For patients treated with lamivudine in study 2301 and enrolled into group B, the total telbivudine treatment time was 104 weeks.

GROUP C: Patients with either compensated or decompensated chronic hepatitis B, who had discontinued study drug treatment in their previous Idenix-sponsored study due to an efficacy response as recommended by protocol. Patients who were eligible for treatment discontinuation in their previous study but who were, at the principal investigators discretion, continued on study therapy, were eligible to enter this study in Group C provided their treatment was discontinued at their last visit of the previous study. The feeder studies for group C of current study were study 2302/015, 2401, 2402, and 010. For patients who enrolled into group C, total telbivudine treatment time was 104 weeks starting from the baseline of the feeder studies to their last visit of the feeder studies. Patients were enrolled to current study (study 2303) for off-treatment follow-up after the treatment discontinuation due to efficacy. Hence, patients did not receive any study drug except in case of patients who relapsed and reinitiated treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient completed a previous qualifying Idenix-Sponsored trial with telbivudine
* Patient was not discontinued from previous Idenix-Sponsored study

Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Patient is pregnant or breastfeeding
* Patient is co-infected with hepatitis C, hepatitis D or HIV

Other protocol-defined exclusion criteria may apply

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1869 (Actual)
Dates: Start 2005-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (18):
  - Novartis Investigational Site, Phoenix, Arizona
  - Novartis Investigational Site, Los Angeles, California
  - Novartis Investigational Site, Pasadena, California
  - Novartis Investigational Site, Sacramento, California
  - Novartis Investigational Site, San Diego, California
  - Novartis Investigational Site, San Francisco, California
  - Novartis Investigational Site, Sarasota, Florida
  - Novartis Investigational Site, Atlanta, Georgia
  - Novartis Investigational Site, Honolulu, Hawaii
  - Novartis Investigational Site, Chicago, Illinois
  - Novartis Investigational Site, Boston, Massachusetts
  - Novartis Investigational Site, Ann Arbor, Michigan
  - Novartis Investigational Site, St Louis, Missouri
  - Novartis Investigational Site, New York, New York
  - Novartis Investigational Site, Chapel Hill, North Carolina
  - Novartis Investigational Site, Philadelphia, Pennsylvania
  - Novartis Investigational Site, Houston, Texas
  - Novartis Investigational Site, Richmond, Virginia
- Novartis Investigational Site, Heidelberg, Victoria, Australia
- Novartis Investigational Site, Toronto, Ontario, Canada
- Novartis Investigational Site, Beijing, Beijing Municipality, China
- Novartis Investigational Site, Prague, Czechia
- Novartis Investigational Site, Paris, France
- Novartis Investigational Site, Hanover, Germany
- Novartis Investigational Site, Hong Kong, Hong Kong
- Novartis Investigational Site, New Delhi, India
- Novartis Investigational Site, Nazareth, Israel
- Novartis Investigational Site, Torino, Italy
- Novartis Investigational Site, Hamilton, New Zealand
- Novartis Investigational Site, Krakow, Poland
- Novartis Investigational Site, Santurce, Puerto Rico
- Novartis Investigational Site, Singapore, Singapore
- Novartis Investigational Site, Seoul, South Korea
- Novartis Investigational Site, Valencia, Spain
- Novartis Investigational Site, Tainan, Taiwan
- Novartis Investigational Site, Bangkok, Thailand
- Novartis Investigational Site, Istanbul, Turkey (Türkiye)
- Novartis Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Hsu CW, Chao YC, Lee CM, Chang TT, Chen YC. Efficacy of telbivudine in Taiwanese chronic hepatitis B patients compared with GLOBE extension study and predicting treatment outcome by HBV DNA kinetics at week 24. BMC Gastroenterol. 2012 Dec 13;12:178. doi: 10.1186/1471-230X-12-178. PMID 23234302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open-label trial of telbivudine in adults with chronic hepatitis B previously treated in Idenix-sponsored telbivudine studies. Study start March 2005 and completed November 2009.
Groups:
- Group A : LdT Pool 2302/015: Subjects with HBeAg (+) or HBeAg (-) compensated chronic hepatitis B from phase III pivotal, registration studies 2302 (NCT00057265) and 015 (NCT00131742) treated with Telbivudine. Telbivudine 600 mg by mouth (p.o.) daily for 104 weeks. The total telbivudine treatment time starting from feeder study baseline to the end of the on-treatment period in study 2303 was 208 weeks.
- Group A : LAM Pool 2302/015: Subjects with HBeAg (+) or HBeAg (-) compensated chronic hepatitis B from phase III pivotal, registration studies 2302 (NCT00057265) and 015 (NCT00131742) treated with Lamivudine. Telbivudine 600 mg by mouth (p.o.) daily for 104 weeks.
- Group A: Feeder Study 2401: Subjects with HBeAg (+) or HBeAg (-) compensated chronic hepatitis B from phase IIIb, registration study CLDT600A2401 (NCT00115245) treated with Telbivudine. Telbivudine 600 mg by mouth (p.o.) daily for 104 weeks.
- Group A: Feeder Study 2402: Subjects with HBeAg (+) or HBeAg (-) compensated chronic hepatitis B from phase IIIb, registration study CLDT600A2402 (NCT00132652) and treated with Lamivudine or Telbivudine. Telbivudine 600 mg by mouth (p.o.) daily for 104 weeks.
- Group A: Feeder Study 010: Subjects with HBeAg (+) or HBeAg (-) compensated chronic hepatitis B were from phase IIb study NV-02B-010 (NCT00124241) of telbivudine, lamivudine or the combination of both agents. Telbivudine 600 mg by mouth (p.o.) daily for 104 weeks.
- Group B: LdT 2301: Subjects with HBeAg (+) or HBeAg (-) decompensated chronic hepatitis B from phase III pivotal, registration study 2301 (NCT00076336) treated with Telbivudine. Telbivudine 600 mg by mouth (p.o.) daily for 104 weeks. The total telbivudine treatment time starting from feeder study baseline to the end of the on-treatment period in study 2303 was 208 weeks.
- Group B: LAM 2301: Subjects with HBeAg (+) or HBeAg (-) decompensated chronic hepatitis B from phase III pivotal, registration studies 2301 (NCT00076336) treated with Lamivudine. Telbivudine 600 mg by mouth (p.o.) daily for 104 weeks.
- Group C: LdT Pool 2302/015: Subjects with either compensated or decompensated chronic hepatitis B from phase III pivotal, registration studies 2302 (NCT00057265) and 015 (NCT00131742) treated with Telbivudine. Patients were enrolled for off-treatment follow-up after the treatment discontinuation due to efficacy at their last visit of the feeder studies. Hence, patients did not receive any study drug except in case of patients who relapsed and reinitiated treatment.
- Group C: LAM Pool 2302/015: Subjects with either compensated or decompensated chronic hepatitis B from phase III pivotal, registration studies 2302 (NCT00057265) and 015 (NCT00131742) treated with Lamivudine. Patients were enrolled for off-treatment follow-up after the treatment discontinuation due to efficacy at their last visit of the feeder studies. Hence, patients did not receive any study drug except in case of patients who relapsed and reinitiated treatment.
- Group C: Other Feeder Studies: Patients with either compensated or decompensated chronic hepatitis B, from 2401 (NCT00115245), 2402 (NCT00132652) and 010 (NCT00124241). Patients were enrolled for off-treatment follow-up after the treatment discontinuation due to efficacy at their last visit of the feeder studies. Hence, patients did not receive any study drug except in case of patients who relapsed and reinitiated treatment.
Period: Overall Study
Arm/Group | Group A : LdT Pool 2302/015 | Group A : LAM Pool 2302/015 | Group A: Feeder Study 2401 | Group A: Feeder Study 2402 | Group A: Feeder Study 010 | Group B: LdT 2301 | Group B: LAM 2301 | Group C: LdT Pool 2302/015 | Group C: LAM Pool 2302/015 | Group C: Other Feeder Studies
Started | 667 | 632 | 123 | 206 | 56 | 26 | 23 | 66 | 57 | 13
Safety Population | 655 | 626 | 122 | 206 | 50 | 26 | 23 | 66 | 57 | 13
Per Protocol Population | 635 | 606 | 120 | 202 | 50 | 25 | 19 | 64 | 56 | 13
Completed | 507 (Completed week 104/week 208.) | 456 | 90 | 121 | 46 | 10 | 15 | 58 | 52 | 13
Not Completed | 160 | 176 | 33 | 85 | 10 | 16 | 8 | 8 | 5 | 0
Not completed — Adverse Event | 10 | 10 | 1 | 5 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Clinical disease progression | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 1 | 1 | 0 | 0 | 6 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 44 | 62 | 9 | 12 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Non-compliance | 15 | 13 | 0 | 6 | 1 | 0 | 0 | 3 | 3 | 0
Not completed — Patient, Investigator,or Sponsor request | 66 | 60 | 11 | 51 | 4 | 3 | 1 | 4 | 1 | 0
Not completed — Pregnancy | 4 | 4 | 2 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Virologic breakthrough | 19 | 23 | 9 | 7 | 2 | 3 | 3 | 0 | 0 | 0
Not completed — Other- not specified | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Treatment Failure | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A : LdT Pool 2302/015: Subjects with HBeAg (+) or HBeAg (-) compensated chronic hepatitis B from phase III pivotal, registration studies Subjects with HBeAg (+) or HBeAg (-) compensated chronic hepatitis B from phase III pivotal, registration studies 2302 (NCT00057265) and 015 (NCT00131742) treated with Telbivudine. Telbivudine 600 mg by mouth (p.o.) daily for 104 weeks. The total telbivudine treatment time starting from feeder study baseline to the end of the on-treatment period in study 2303 was 208 weeks.
- Total: Total of all reporting groups
Arm/Group | Group A : LdT Pool 2302/015 | Group A : LAM Pool 2302/015 | Group A: Feeder Study 2401 | Group A: Feeder Study 2402 | Group A: Feeder Study 010 | Group B: LdT 2301 | Group B: LAM 2301 | Group C: LdT Pool 2302/015 | Group C: LAM Pool 2302/015 | Group C: Other Feeder Studies | Total
Number analyzed (Participants) | 667 | 632 | 123 | 206 | 56 | 26 | 23 | 66 | 57 | 13 | 1869
Age, Customized [Number; unit: Participants]
  < 30 years | 276 | 207 | 51 | 54 | 9 | 1 | 0 | 30 | 27 | 8 | 663
  30-50 years | 320 | 325 | 66 | 122 | 40 | 10 | 5 | 31 | 24 | 5 | 948
  > 50 years | 71 | 100 | 6 | 30 | 7 | 15 | 18 | 5 | 6 | 0 | 258
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 142 | 30 | 53 | 9 | 9 | 6 | 20 | 14 | 3 | 433
  Male | 520 | 490 | 93 | 153 | 47 | 17 | 17 | 46 | 43 | 10 | 1436

OUTCOME MEASURES:

1. Secondary Outcome: To Longitudinally Assess the Longer-term Antiviral Efficacy Achieved With Telbivudine Treatment
Time Frame: 52 weeks, 104 weeks, 156 weeks, 208 weeks
Reporting Status: Not Posted

2. Secondary Outcome: To Longitudinally Assess the Clinical Efficacy of Longer-term Treatment With Telbivudine
Time Frame: 52 weeks, 104 weeks, 156 weeks, 208 weeks
Reporting Status: Not Posted

3. Secondary Outcome: To Longitudinally Assess the Durability of HBeAg Responses Achieved With Telbivudine Treatment and Other Previous Treatments in Patients
Time Frame: 52 weeks, 104 weeks, 156 weeks, 208 weeks
Reporting Status: Not Posted

4. Secondary Outcome: To Determine the Longitudinal Frequency of Virologic Breakthrough and Characterize the Associated Mutations in the HBV Polymerase Gene in HBV DNA Amplified From Sera of Patients With Virologic Breakthrough
Time Frame: 52 weeks, 104 weeks, 156 weeks, 208 weeks
Reporting Status: Not Posted

5. Primary Outcome: Percentage of Participants Who Maintained Therapeutic Response [Group A: LdT Pool 2302/015]
Description: The maintained therapeutic response is defined as hepatitis B virus (HBV) DNA < 5 log10 copies/mL and either hepatitis Be antigen (HBeAg) loss or alanine aminotransferase (ALT) normalized. HBeAg loss is loss of detectable serum HBeAg in a patient who was HBeAg-positive at feeder baseline. ALT normalized is defined as ALT within normal limits for a patient with an elevated ALT level (>1.0 × ULN) at either the feeder baseline or feeder screening visit. All efficacy data were analyzed separately for HBeAg-positive and HBeAg-negative patients.
Time Frame: 156 weeks, 208 weeks (from feeder study baseline)
Population: Per protocol (PP) population. The PP analysis was done on separately for the HBeAg-positive and HBeAg-negative subpopulation (status at feeder baseline). n = the number of HBeAg-positive/HBeAg-negative patients who were eligible for maintained therapeutic response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A : LdT Pool 2302/015
Number analyzed (Participants) | 635
Percentage of participants
  HBeAg Positive: week 156 (n=338) | 67.2 [61.9 to 72.1]
  HBeAg Positive: week 208 (n=252) | 73.8 [67.9 to 79.1]
  HBeAg Negative: week 156 (n=197) | 81.7 [75.6 to 86.9]
  HBeAg Negative: week 208 (n=168) | 86.3 [80.2 to 91.1]

6. Primary Outcome: Percentage of Participants Who Maintained Therapeutic Response [Group A: LAM Pool 2302/015]
Description: as for outcome 5
Time Frame: 52 weeks, 104 weeks
Population: Per protocol (PP) population. The PP analysis was done separately for the HBeAg-positive and HBeAg-negative subpopulation (status at feeder baseline). n = the number of HBeAg-positive/HBeAg-negative patients who were eligible for maintained therapeutic response.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group A : LAM Pool 2302/015
Number analyzed (Participants) | 606
Percentage of Participants
  HBeAg Positive: week 52 (n=338) | 60.1 [54.6 to 65.3]
  HBeAg Positive: week 104 (n=101) | 65.3 [55.2 to 74.5]
  HBeAg Negative: week 52 (n=182) | 80.8 [74.3 to 86.2]
  HBeAg Negative: week 104 (n=79) | 81.0 [70.6 to 89.0]

7. Primary Outcome: Percentage of Participants Who Maintained Therapeutic Response [Group A: Feeder Studies 2401/2402/010]
Description: as for outcome 5
Time Frame: 52 weeks, 104 weeks
Population: Per protocol (PP) population. The PP analysis was done on the PP population, separately for the HBeAg-positive and HBeAg-negative subpopulation (status as feeder baseline). n = the number of HBeAg-positive/HBeAg-negative patients who were eligible for maintained therapeutic response.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group A: Feeder Study 2401 | Group A: Feeder Study 2402 | Group A: Feeder Study 010
Number analyzed (Participants) | 120 | 131 | 50
Percentage of Participants
  HBeAg Positive: 52 week (n = 103, 79, 43) | 77.7 [68.4 to 85.3] | 35.4 [25.0 to 47.0] | 69.8 [53.9 to 82.8]
  HBeAg Positive: 104 week (n = 66, 15, 30) | 81.8 [70.4 to 90.2] | 46.7 [21.3 to 73.4] | 76.7 [57.7 to 90.1]
  HBeAg Negative: 52 week (n = 0, 37, 0) | NA [NA to NA] — In per protocol population, all participants from feeder study 2401 are HBeAg-positive. So, no analysis was done at week 52. | 54.1 [36.9 to 70.5] | NA [NA to NA] — In per protocol population, all participants from feeder study 010 are HBeAg-positive. So, no analysis was done at week 52.
  HBeAg Negative: 104 week (n = 0, 10, 0) | NA [NA to NA] — In per protocol population, all participants from feeder study 2401 are HBeAg-positive. So, no analysis was done at week 104. | 60.0 [26.2 to 87.8] | NA [NA to NA] — In per protocol population, all participants from feeder study 010 are HBeAg-positive. So, no analysis was done at week 104.

8. Primary Outcome: Percentage of Participants With Maintained Clinical Response [Group B: LdT 2301]
Description: Maintained clinical response is defined as achievement of serum HBV DNA < 4 log10 copies/mL, normal serum ALT level and improvement or stabilization in Child-Turcotte-Pugh (CTP) score. Total CTP score ranges from 5 to 15; higher scores indicate liver impairment. Improvement is defined as a 2-point or greater reduction in CTP score, and stabilization is defined as a less than 2-point change in CTP score, compared to the patient's baseline value. Analysis was done on the overall per protocol (PP) population and separately for the HBeAg-positive and HBeAg-negative subpopulation.
Time Frame: 156 weeks, 208 weeks (from feeder study baseline)
Population: Per protocol (PP) population. The PP analysis was done on the overall PP population and separately for the HBeAg-positive and HBeAg-negative subpopulation (status at feeder baseline). n = the number of patients who were eligible for maintained clinical response.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Group B : LdT 2301: Subjects with HBeAg (+) or HBeAg (-) decompensated chronic hepatitis B from phase III pivotal, registration study 2301 (NCT00076336) treated with Telbivudine. Telbivudine 600 mg by mouth (p.o.) daily for 104 weeks. The total telbivudine treatment time starting from feeder study baseline to the end of the on-treatment period in study 2303 was 208 weeks.
Arm/Group | Group B : LdT 2301
Number analyzed (Participants) | 25
Percentage of Participants
  HBeAg Positive: week 156 (n= 4) | 100 [39.8 to 100]
  HBeAg Positive: week 208 (n= 1) | 100 [2.5 to 100]
  HBeAg Negative: week 156 (n= 11) | 72.7 [39.0 to 94.0]
  HBeAg Negative: week 208 (n= 7) | 71.4 [29.0 to 96.3]
  Overall: Week 156 (n= 15) | 80.0 [51.9 to 95.7]
  Overall: Week 208 (n= 8) | 75.0 [34.9 to 96.8]

9. Primary Outcome: Percentage of Participants With Maintained Clinical Response [Group B: LAM 2301]
Description: as for outcome 8
Time Frame: 52 weeks,104 weeks
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Group B : LAM 2301: Subjects with HBeAg (+) or HBeAg (-) decompensated chronic hepatitis B from phase III pivotal, registration studies 2301 (NCT00076336) treated with Lamivudine. Telbivudine 600 mg by mouth (p.o.) daily for 104 weeks.
Arm/Group | Group B : LAM 2301
Number analyzed (Participants) | 19
Percentage of Participants
  HBeAg Positive: week 52 (n=4) | 100 [39.8 to 100]
  HBeAg Positive: week 104 (n=1) | 100 [2.5 to 100]
  HBeAg Negative: week 52 (n=11) | 72.7 [39.9 to 94]
  HBeAg Negative: week 104 (n=5) | 100 [47.8 to 100]
  Overall: week 52 (n= 15) | 80.0 [51.9 to 95.7]
  Overall: week 104 (n= 6) | 100 [54.1 to 100]

10. Primary Outcome: Percentage of Participants With Sustained Therapeutic Response [Group C: LdT Pool and LAM Pool (2302/015)]
Description: The primary efficacy endpoint for Group C patients was the percentage of patients with sustained therapeutic response (defined as HBV DNA < 5 log10 copies/mL and either HBeAg loss or ALT normalized) at Weeks 52 and 104 of off-treatment follow-up. HBeAg loss is loss of detectable serum HBeAg in a patient who was HBeAg-positive at feeder baseline. ALT normalized is ALT within normal limits for a patient with an elevated ALT level (>1.0 × ULN) at either the feeder baseline or feeder screening visit. All efficacy data were analyzed separately for HBeAg-positive and HBeAg-negative patients.
Time Frame: 52 weeks,104 weeks
Population: The per protocol population. n= is the number of HBeAg-positive/HBeAg-negative patients from per protocol population who achieved maintained response at the end of treatment and had off-treatment assessment to determine the sustained response at that time point or lost sustained response before the off-treatment timepoint.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Group C : LdT Pool 2302/015: Subjects with either compensated or decompensated chronic hepatitis B from phase III pivotal, registration studies 2302 (NCT00057265) and 015 (NCT00131742) treated with Telbivudine. Patients were enrolled for off-treatment follow-up after the treatment discontinuation due to efficacy at their last visit of the feeder studies. Hence, patients did not receive any study drug except in case of patients who relapsed and reinitiated treatment.
Arm/Group | Group C : LdT Pool 2302/015 | Group C: LAM Pool 2302/015
Number analyzed (Participants) | 64 | 56
Percentage of Participants
  HBeAg Positive: week 52 (n= 53, 42) | 69.8 [55.7 to 81.7] | 73.8 [58.0 to 86.1]
  HBeAg Positive: week 104 (n= 42, 32) | 57.1 [41.0 to 72.3] | 62.5 [43.7 to 78.9]
  HBeAg Negative: week 52 (n= 3, 5) | 0.0 [0.0 to 70.8] | 80.0 [28.4 to 99.5]
  HBeAg Negative: week 104 (n= 3, 6) | 0.0 [0.0 to 70.8] | 83.3 [35.9 to 99.6]

11. Primary Outcome: Percentage of Participants With Sustained Therapeutic Response [Group C: Other Feeder Studies]
Description: The primary efficacy endpoint for Group C (other feeder studies) was the percentage of patients with sustained therapeutic response (defined as HBV DNA < 5 log10 copies/mL and either HBeAg loss or ALT normalized) at Weeks 52 and 104 of off-treatment follow-up.
  Patients were enrolled for off-treatment follow-up after the treatment discontinuation due to efficacy at their last visit of the feeder studies. Hence, patients did not receive study drug except in case of patients who relapsed and reinitiated treatment. No statistical summary was performed , only patient listing was generated.
Time Frame: 52 weeks,104 weeks
Population: In "Group C: other feeder study" reporting group, there were only 13 patients; hence, no summary statistics were performed. Only listings were generated.
Groups:
- Group C : Other Feeder Studies: Patients with either compensated or decompensated chronic hepatitis B, from 2401 (NCT00115245), 2402 (NCT00132652) and 010 (NCT00124241). Patients were enrolled for off-treatment follow-up after the treatment discontinuation due to efficacy at their last visit of the feeder studies. Hence, patients did not receive any study drug except in case of patients who relapsed and reinitiated treatment.
Arm/Group | Group C : Other Feeder Studies
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: All safety analyses were performed on the safety populations defined for each reporting group.
Groups:
- Group A: Feeder 2401: Subjects with HBeAg (+) or HBeAg (-) compensated chronic hepatitis B from phase IIIb, registration study CLDT600A2401 (NCT00115245) treated with Telbivudine. Telbivudine 600 mg by mouth (p.o.) daily for 104 weeks.
- Group A: Feeder 2402: Subjects with HBeAg (+) or HBeAg (-) compensated chronic hepatitis B from phase IIIb, registration study CLDT600A2402 (NCT00132652) and treated with Lamivudine or Telbivudine. Telbivudine 600 mg by mouth (p.o.) daily for 104 weeks.
Arm/Group | Group A : LdT Pool 2302/015 | Group A : LAM Pool 2302/015 | Group A: Feeder Study 010 | Group A: Feeder 2401 | Group A: Feeder 2402 | Group B: LdT 2301 | Group B: Lam 2301 | Group C : LdT Pool 2302/015 | Group C: Lam Pool 2302/015 | Group C : Other Feeder Studies
Serious Adverse Events (participants affected / at risk) | 45/655 | 21/626 | 3/50 | 10/122 | 14/206 | 16/26 | 10/23 | 1/66 | 2/57 | 2/13
Other Adverse Events (participants affected / at risk) | 318/655 | 309/626 | 24/50 | 74/122 | 88/206 | 21/26 | 19/23 | 40/66 | 33/57 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A : LdT Pool 2302/015 (N=655) | Group A : LAM Pool 2302/015 (N=626) | Group A: Feeder Study 010 (N=50) | Group A: Feeder 2401 (N=122) | Group A: Feeder 2402 (N=206) | Group B: LdT 2301 (N=26) | Group B: Lam 2301 (N=23) | Group C : LdT Pool 2302/015 (N=66) | Group C: Lam Pool 2302/015 (N=57) | Group C : Other Feeder Studies (N=13)
APLASIA PURE RED CELL (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ANGINA PECTORIS (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VESTIBULAR NEURONITIS (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
ASCITES (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ENTERITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MELAENA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OESOPHAGEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PERITONEAL ADHESIONS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
APLASIA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
CONCOMITANT DISEASE PROGRESSION (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
DEATH (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CHRONIC HEPATITIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEPATITIS (Hepatobiliary disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEPATOMEGALY (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
APPENDICITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DENGUE FEVER (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DENTAL CARIES (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
EPIGLOTTITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HEPATITIS B (Infections and infestations) | 3 | 5 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
LEPTOSPIROSIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PERITONITIS BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PHARYNGITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
POSTOPERATIVE INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SEPTIC SHOCK (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SINUSITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
UROSEPSIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
JOINT LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
JOINT SPRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TOOTH INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 4 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
WEIGHT DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DIABETIC HYPEROSMOLAR NON-KETOACIDOSIS (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
MUSCLE ATROPHY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
POLYMYOSITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ACOUSTIC NEUROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1 | 0 | 0 | 1 | 8 | 3 | 0 | 0 | 0
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
NASAL NEOPLASM BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
POLYP (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PROLACTINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RENAL CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
THYROID GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DIABETIC HYPEROSMOLAR COMA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ABORTION (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABORTION MISSED (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ADJUSTMENT DISORDER (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPOMANIA (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
CALCULUS URINARY (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GLOMERULONEPHRITIS PROLIFERATIVE (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
OBSTRUCTIVE UROPATHY (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PROTEINURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
METRORRHAGIA (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PROSTATIC HYPERTROPHY (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
VULVAL ANGIOKERATOMA (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CATARRH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NASAL MUCOSAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NASAL TURBINATE ABNORMALITY (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ABORTION INDUCED (Surgical and medical procedures) | 4 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
FRACTURE TREATMENT (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLEEDING VARICOSE VEIN (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A : LdT Pool 2302/015 (N=655) | Group A : LAM Pool 2302/015 (N=626) | Group A: Feeder Study 010 (N=50) | Group A: Feeder 2401 (N=122) | Group A: Feeder 2402 (N=206) | Group B: LdT 2301 (N=26) | Group B: Lam 2301 (N=23) | Group C : LdT Pool 2302/015 (N=66) | Group C: Lam Pool 2302/015 (N=57) | Group C : Other Feeder Studies (N=13)
THROMBOCYTHAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 10 | 13 | 1 | 2 | 1 | 1 | 2 | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 8 | 10 | 1 | 2 | 8 | 1 | 3 | 1 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 26 | 15 | 3 | 5 | 5 | 3 | 3 | 3 | 2 | 0
ABDOMINAL SYMPTOM (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
ASCITES (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 11 | 8 | 3 | 1 | 1 | 0 | 2 | 1 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 21 | 21 | 2 | 1 | 2 | 1 | 4 | 3 | 2 | 0
DYSPEPSIA (Gastrointestinal disorders) | 12 | 12 | 1 | 4 | 2 | 2 | 0 | 2 | 2 | 1
GINGIVAL BLEEDING (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 10 | 18 | 2 | 3 | 2 | 3 | 1 | 1 | 1 | 1
VOMITING (Gastrointestinal disorders) | 6 | 9 | 2 | 1 | 1 | 1 | 2 | 0 | 0 | 1
ASTHENIA (General disorders) | 9 | 6 | 0 | 6 | 4 | 0 | 2 | 1 | 1 | 0
FATIGUE (General disorders) | 29 | 33 | 2 | 7 | 5 | 0 | 5 | 12 | 3 | 3
MALAISE (General disorders) | 2 | 2 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 4 | 4 | 0 | 0 | 1 | 4 | 4 | 0 | 0 | 0
PITTING OEDEMA (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
PYREXIA (General disorders) | 11 | 11 | 1 | 2 | 4 | 4 | 1 | 2 | 0 | 1
HEPATIC LESION (Hepatobiliary disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 | 7 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1
HYPERSENSITIVITY (Immune system disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
BODY TINEA (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 5 | 5 | 1 | 2 | 2 | 2 | 0 | 1 | 0 | 0
HEPATITIS B (Infections and infestations) | 16 | 7 | 3 | 2 | 9 | 1 | 1 | 2 | 1 | 1
INFLUENZA (Infections and infestations) | 25 | 22 | 11 | 6 | 1 | 1 | 0 | 4 | 3 | 1
NASOPHARYNGITIS (Infections and infestations) | 69 | 73 | 1 | 18 | 6 | 1 | 3 | 2 | 1 | 1
TINEA VERSICOLOUR (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
TONSILLITIS (Infections and infestations) | 4 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 50 | 60 | 2 | 24 | 9 | 4 | 4 | 15 | 14 | 1
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 0
JOINT SPRAIN (Injury, poisoning and procedural complications) | 4 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
POST PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 4 | 1 | 0 | 2 | 0 | 0 | 2 | 1 | 1 | 0
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 18 | 12 | 1 | 0 | 9 | 0 | 0 | 0 | 1 | 2
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 56 | 47 | 2 | 5 | 24 | 3 | 4 | 2 | 0 | 2
HBV DNA INCREASED (Investigations) | 1 | 1 | 0 | 0 | 12 | 0 | 0 | 0 | 1 | 1
WEIGHT DECREASED (Investigations) | 3 | 4 | 0 | 1 | 3 | 1 | 2 | 0 | 0 | 0
WEIGHT INCREASED (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
DIABETES MELLITUS NON-INSULIN-DEPENDENT (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 18 | 15 | 1 | 4 | 6 | 1 | 3 | 1 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 16 | 16 | 1 | 2 | 8 | 1 | 2 | 3 | 2 | 2
MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 8 | 10 | 0 | 2 | 2 | 2 | 1 | 1 | 3 | 0
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
DIZZINESS (Nervous system disorders) | 7 | 7 | 1 | 4 | 4 | 2 | 1 | 2 | 0 | 1
HEADACHE (Nervous system disorders) | 28 | 28 | 2 | 5 | 9 | 2 | 2 | 2 | 1 | 2
DEPRESSION (Psychiatric disorders) | 5 | 4 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
GLOMERULONEPHRITIS PROLIFERATIVE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 27 | 22 | 1 | 4 | 12 | 3 | 2 | 3 | 4 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 17 | 11 | 1 | 7 | 5 | 1 | 0 | 3 | 1 | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0 | 3 | 2 | 0 | 2 | 0 | 1 | 0
ACNE (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 3 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1
PALMAR ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 12 | 6 | 0 | 7 | 2 | 2 | 0 | 2 | 0 | 2
SPIDER NAEVUS (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
EYE OPERATION (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPERTENSION (Vascular disorders) | 11 | 15 | 0 | 5 | 1 | 1 | 2 | 0 | 0 | 1
VARICOSE VEIN (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial; or the publication of the trial results in their entirety.